CLINICAL TRIAL: NCT03943914
Title: Early Non-invasive Ventilation and High-flow Nasal Oxygen Therapy for Preventing Delayed Respiratory Failure in Hypoxemic Blunt Chest Trauma Patients.
Acronym: OptiTHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2018/62
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Chest Injuries; Respiratory Failure
Keywords: Chest trauma; Respiratory failure; Noninvasive ventilation; High-flow nasal oxygen therapy
MeSH Terms: conditions — Thoracic Injuries; Respiratory Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An "early" NIV strategy associated with HFNC-O2 (Experimental)
  Interventions: Combination Product: Preventive strategy
- A "late" NIV strategy associated with COT (Active Comparator)
  Interventions: Combination Product: Standard of care

INTERVENTIONS:
Combination Product: Preventive strategy — In the experimental strategy, NIV is performed after inclusion in patients with moderate hypoxemia, defined by a PaO2/FiO2 ratio < 300 mmHg. The minimally required duration of NIV was 4 hours per day for at least 2 calendar days. The daily duration of NIV can be increased at the discretion of the physician in patients with signs of delayed respiratory failure under HFNC-O2 and improving under NIV. Beyond the first 48 hours, NIV and HFNC-O2 can be stopped and the patient switched to COT if respiratory rate < 25/min and SpO2 > 92% under FiO2 < 30% for at least 6 hours.
  Arms: An "early" NIV strategy associated with HFNC-O2
Combination Product: Standard of care — In the control group, patients receive oxygen from nasal cannula or high concentration oxygen mask according to the FiO2 needed to achieve SpO2 > 92%. NIV is initiated only in patients having PaO2/FiO2 ratio < 200 mmHg under COT. A trial of curative NIV is allowed at the discretion of the physician in patients who have signs of delayed respiratory failure and no other organ dysfunction. The non-improvement of respiratory conditions after 1 hour of NIV, the NIV-dependence (≥ 12 consecutive hours) or NIV-intolerance should be considered as criteria for endotracheal intubation.
  Arms: A "late" NIV strategy associated with COT

SUMMARY:
In blunt chest trauma patients without immediate life-threatening conditions, delayed respiratory failure and need for mechanical ventilation may still occur in 12 to 40% of patients, depending on the severity of the trauma, the preexisting conditions and the intensity of initial management.

In this context, non-invasive ventilation (NIV) is recommended in hypoxemic chest trauma patients, defined as a PaO2/FiO2 ratio < 200 mmHg. However, there is a large heterogeneity among studies regarding the severity of injuries, the degree of hypoxemia and the timing of enrollment. The interest of a preventive strategy during the early phase of blunt chest trauma, before the occurrence of respiratory distress or severe hypoxemia, is not formally established in the literature. Moreover, high-flow nasal oxygen therapy (HFNC-O2) appears to be a reliable and better tolerated alternative to conventional oxygen therapy (COT), associated with a significant reduction in intubation rate in hypoxemic patients.

Two NIV strategies are compared:

1. In the experimental strategy, NIV is performed after inclusion in patients with moderate hypoxemia, defined by a PaO2/FiO2 ratio < 300 mmHg. The minimally required duration of NIV was 4 hours per day for at least 2 calendar days.
2. In the control group, patients receive oxygen from nasal cannula or high concentration oxygen mask according to the FiO2 needed to achieve SpO2 > 92%. NIV is initiated only in patients having PaO2/FiO2 ratio < 200 mmHg under COT.

Investigators hypothesized that an early strategy associating HFNC-O2 and preventive NIV in hypoxemic blunt chest trauma patients may reduce the need for mechanical ventilation compared to the recommended strategy associating COT and late NIV.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in intensive care unit within 48 hours after a high-risk blunt chest trauma, defined by a TTS (Thorax Trauma Severity) score ≥ 8.
* Hypoxemia defined by a PaO2/FiO2 ratio < 300, and the absence of hypercapnia (PaCO2 < 45 mmHg).
* Without indication of endotracheal intubation at inclusion.
* Affiliated person or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Criteria relating to formal indication to NIV: Exacerbation of underlying chronic respiratory disease, cardiogenic pulmonary edema, severe neutropenia.
* Criteria relating to contraindications to NIV: Hemodynamic instability, Glasgow Coma Scale score ≤ 12 or excessive agitation, or other contraindications to non-invasive ventilation (active gastrointestinal bleeding, low level of consciousness, multiorgan failure, airway patency problems, lack of cooperation or hemodynamic instability).
* Associated traumatic lesions entailing particular risks: severe brain injury, complex facial trauma, tetraplegia, tracheobronchial or esophageal injuries, thoracic or abdominal trauma with indication for surgery by thoracotomy or laparotomy.
* Criteria relating to the regulation: A do-not-intubate order and a decision not to participate, persons placed under judicial protection, persons participating in another research including a period of exclusion still in course, severely altered physical and/or psychological health which, according to the investigator, could affect the participant's compliance of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Necessity to perform endotracheal intubation | Up to 14 days after randomization
  To ensure the consistency of indications across sites and reduce the risk of delayed intubation, the following criteria for endotracheal intubation must be used (only one criterion is needed): cardiac arrest or significant hemodynamic instability, deterioration of neurologic status, signs of persisting or worsening respiratory failure as defined by at least two of the following criteria: respiratory rate of more than 35 breaths per minute, lack of improvement in signs of high respiratory-muscle workload, development of copious tracheal secretions, signs of respiratory exhaustion (pH <7.32 or PaCO2 > 50 mmHg), major hypoxemia (PaO2/FiO2 ratio <100 or SpO2 <92% for more than 5 minutes).

SECONDARY OUTCOMES:
PaO2/FiO2 ratio | every 6 hours during the first 48 hours after randomization
Respiratory rate | every 6 hours during the first 48 hours after randomization
Dyspnea score | every 6 hours during the first 48 hours after randomization
  Dyspnea score : +2 = significant improvement; +1 = slight improvement; 0 = no change; -1 = slight deterioration ; -2 = significant deterioration
ICU and hospital length of stay | Up to 14 days after randomization
ICU or in-hospital mortality | Up to 14 days after randomization
Number of ventilator free-days | Up to 14 days after randomization
  Days alive and without invasive or non-invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche Clinique et Epidémiologique (USMR) du CHU de Bordeaux
Locations (14):
- France (14):
  - CHU Amiens-Picardie, Amiens
  - CH d'Annecy, Annecy
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - APHP - Hôpital Beaujon, Clichy
  - AP-HM - Hôpital de la Timone, Marseille
  - CHU de Nîmes, Nîmes
  - CH de Pau, Pau
  - HCL - Hôpital Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
  - CHU de Strasbourg - Hôpital Civil, Strasbourg
  - CHU de Strasbourg -Hôpital de Hautepierre, Strasbourg
  - Hôpital Robert Picqué, Villenave-d'Ornon

IPD SHARING:
Plan to Share IPD: No